CLINICAL TRIAL: NCT00412594
Title: Phase II Study of 2-Chlorodeoxyadenosine (2CDA) Followed by Rituximab in Hairy Cell Leukemia
Brief Title: Cladribine and Rituximab in Treating Patients With Hairy Cell Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0223; NCI-2012-01394 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2004-0223 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2006-12-14; First posted 2006-12-18 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Hairy Cell Leukemia; Recurrent Hairy Cell Leukemia
MeSH Terms: conditions — Leukemia, Hairy Cell | interventions — Cladribine; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cladribine and rituximab) (Experimental): Patients receive cladribine IV over 2 hours QD on days 1-5 and rituximab IV once weekly for 8 weeks beginning on day 28 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cladribine; Other: Laboratory Biomarker Analysis; Biological: Rituximab

INTERVENTIONS:
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima

SUMMARY:
This phase II trial studies the side effects and how well cladribine and rituximab work in treating patients with hairy cell leukemia. Drugs used in chemotherapy, such as cladribine, work in different ways to stop the growth of cancer cells either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as rituximab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving cladribine together with rituximab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate the efficacy in achieving complete response of combination of cladribine administered intravenously over 2 hours for 5 days followed by rituximab weekly for 8 weeks in patients with untreated or previously treated hairy cell leukemia.

II. To examine the efficacy of rituximab to eradicate minimal residual disease (MRD) after cladribine therapy (as assessed by immunophenotyping of bone marrow and peripheral blood).

III. To examine the effect of addition of rituximab to cladribine on the long term disease-free (DFS) and overall survival (OS) (as compared with historical controls).

IV. To evaluate potential predictors of outcome including molecular and flow evaluations of MRD, as well as other potential molecular predictors such as v-raf murine sarcoma viral oncogene homolog B1 (BRAF).

OUTLINE:

Patients receive cladribine intravenously (IV) over 2 hours once daily (QD) on days 1-5 and rituximab IV once weekly for 8 weeks beginning on day 28 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of hairy cell leukemia (HCL) established by bone marrow examination
* Patients with relapsed disease are eligible if they have had no more than one prior therapy
* Women of child-bearing potential must use birth control (oral contraceptive, barrier, abstinence or any other acceptable method) for the duration of the study
* Performance status =< 3
* Creatinine less than or equal to 2.0 unless related to the disease
* Bilirubin less than or equal to 3.0
* Transaminases less than or equal 3 x upper limit of normal unless related to the disease
* No prior investigational agent in the 4 weeks prior to initiation of therapy

Exclusion Criteria:

* Unable or unwilling to sign the consent form
* Known infection with human immunodeficiency virus (HIV), hepatitis B or C
* Presence of active infection
* Presence of central nervous system (CNS) metastases
* New York Heart Association classification III or IV heart disease
* Prior chemotherapy (last 4 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2004-06-10 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of rituximab on achievement of complete response after therapy with cladribine | At 12 weeks
  Defined as the absence of hairy cells in the bone marrow or the presence of less than 1 percent atypical cells and the disappearance of all evidence of hairy cell leukemia on physical examination. Monitored using the method of Thall, Simon, Estey as extended by Thall and Sung.
Monitoring the related toxicity for the therapy Grade 3-4 | Up to 1 year
  Monitored using the method of Thall, Simon, Estey as extended by Thall and Sung.
Efficacy of rituximab in eradication of minimal residual disease after cladribine therapy, assessed by immunophenotyping of bone marrow and peripheral blood | Up to 4 weeks after the last dose of rituximab
  The method of Thall, Simon, Estey as extended by Thall and Sung will be used for efficacy and safety monitoring.
Efficacy of rituximab on prolongation of event-free survival | Up to 1 year
Efficacy of rituximab on prolongation of overall survival | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ravandi F, O'Brien S, Jorgensen J, Pierce S, Faderl S, Ferrajoli A, Koller C, Challagundla P, York S, Brandt M, Luthra R, Burger J, Thomas D, Keating M, Kantarjian H. Phase 2 study of cladribine followed by rituximab in patients with hairy cell leukemia. Blood. 2011 Oct 6;118(14):3818-23. doi: 10.1182/blood-2011-04-351502. Epub 2011 Aug 5. PMID 21821712
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org